CLINICAL TRIAL: NCT05800886
Title: The Effect of Early Mobilization With Tea, Coffee and Warm Water Consumption on Bowel Movements in Patients Undergoing Laparoscopic Cholecystectomy Surgery
Brief Title: The Effect of Early Mobilization and Fluid Consumption on Bowel Movements After Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Burçin IRMAK, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GaziU-SBF-BI-1
Record Dates: First submitted 2023-03-12; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Cholelithiases; Nursing Caries; Perioperative Complication; Bowel Ileus
Keywords: Laparoscopic cholecystectomy; Early mobilization; Tea; Coffee; Water consumption; Intestines; Nursing
MeSH Terms: conditions — Cholelithiasis; Ileus | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tea Group (Experimental): At the 4th hour postoperatively, the patients in the tea group were first mobilized after drinking 200 ml of tea within 15 minutes. Patients were supported by the investigator for early mobilization from the 4th hour after surgery.
  Interventions: Other: Early mobilization and tea consumption
- Coffee Group (Experimental): At the 4th hour postoperatively, the patients in the tea group were first mobilized after drinking 200 ml of coffee within 15 minutes. Patients were supported by the investigator for early mobilization from the 4th hour after surgery.
  Interventions: Other: Early mobilization and coffee consumption
- Warm Water Group (Experimental): At the 4th hour postoperatively, the patients in the tea group were first mobilized after drinking 200 ml of warm water within 15 minutes. Patients were supported by the investigator for early mobilization from the 4th hour after surgery.
  Interventions: Other: Early mobilization and warm water consumption
- Control Group (Active Comparator): The first mobilization and oral intake of the patients in the control group started at the 8th hour. Control group didn't receive any intervention. Participants received usual care from health professionals.
  Interventions: Other: Ongoing treatment

INTERVENTIONS:
Other: Early mobilization and tea consumption — At the 4th hour postoperatively, the patients in the tea group were first mobilized after drinking 200 ml of tea (black tea 2 g, caffeine amount: 45-55 mg/150 ml) within 15 minutes. A thermos cup is used to prevent the heat loss of the beverage. Patients were supported by the investigator for early mobilization from the 4th hour after surgery. After the surgery, the first mobilization of the patients is in the form of walking in the patient room of 10 meters (5 meters going and 5 meters returning). According to Enhanced Recovery After Surgery protocols, it is aimed for the patient to walk for at least 2 hours after surgery.
  Arms: Tea Group
Other: Early mobilization and coffee consumption — At the 4th hour postoperatively, the patients in the tea group were first mobilized after drinking 200 ml of coffee (ınstant coffee 2 g, caffeine amount: 60/80 mg/150 ml) within 15 minutes. A thermos cup is used to prevent the heat loss of the beverage. Patients were supported by the investigator for early mobilization from the 4th hour after surgery. After the surgery, the first mobilization of the patients is in the form of walking in the patient room of 10 meters (5 meters going and 5 meters returning). According to Enhanced Recovery After Surgery protocols, it is aimed for the patient to walk for at least 2 hours after surgery.
  Arms: Coffee Group
Other: Early mobilization and warm water consumption — At the 4th hour postoperatively, the patients in the tea group were first mobilized after drinking 200 ml of warm water (37 centigrade) within 15 minutes. A thermos cup is used to prevent the heat loss of the beverage. Patients were supported by the investigator for early mobilization from the 4th hour after surgery. After the surgery, the first mobilization of the patients is in the form of walking in the patient room of 10 meters (5 meters going and 5 meters returning). According to Enhanced Recovery After Surgery protocols, it is aimed for the patient to walk for at least 2 hours after surgery.
  Arms: Warm Water Group
Other: Ongoing treatment — The first mobilization and oral intake of the patients in the control group started at the 8th hour.
  Arms: Control Group

SUMMARY:
Objective: The aim of this study was to determine the effect of early mobilization with consumption of tea, coffee, and warm water on bowel movements in patients who had laparoscopic cholecystectomy surgery.

Design: The study was a single-center, parallel, randomized, controlled trial. Setting: This study was carried out in the general surgery clinic of a university hospital in Türkiye.

Metod: The participants were randomized into four equal groups: tea, coffee, arm water and control. At the 4th hour postoperatively, the patients in the intervention group were first mobilized after drinking 200 ml of tea, coffee or warm water within 15 minutes. The first mobilization and oral intake of the patients in the control group started at the 8th hour. Bowel movements, mobilization time, first flatulence, first stool removal and hospital stay of the patients were followed up. Data were collected with "Patient Information Form", "Glasgow Coma Scale", "Patient Mobilization Follow-up Form" and "Patient Undergone Laparoscopic Cholecystectomy Surgery Follow-Up Form".

Hypothesis:

H0-a: Early mobilization and tea consumption have no effect on the first flatulence time in patients who have undergone laparoscopic cholecystectomy surgery.

H0-b: Early mobilization and coffee consumption have no effect on the first flatulence time in patients who have undergone laparoscopic cholecystectomy.

H0-c: Early mobilization and consumption of warm water have no effect on the initial flatulence time in patients who have undergone laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the study
* To be the age is between 18 and 65 years old
* To undergone laparoscopic cholecystectomy surgery
* To have American Society of Anesthesiologists (ASA) classification I or II

Exclusion Criteria:

* To have a history of cesarean section, hysterectomy, extensive intra-abdominal surgery
* To have metastatic disease, inflammatory bowel disease
* To use drugs that may affect intestinal functions due to systemic diseases
* To known allergy or sensitivity to coffee/caffeine
* To having difficulty swallowing
* To have mental disability or perception problems
* To have a barrier to communication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
First flatus time | up to 24 hours after surgery
  The patient's first flatus output time was questioned. The hour reported by the patient was evaluated as the time of first flatus.

SECONDARY OUTCOMES:
Mobilization time | up to 24 hours after surgery
  The duration of mobilization for the first 24 hours after surgery were evaluated with Patient Mobilization Follow-up Form.
First defecation time | up to 24 hours after surgery
  The patient's first defecation time was questioned. The hour reported by the patient was evaluated as the time of first defecation.
Bowel movements | up to 8 hours after surgery
  Bowel movements were listened to with the same stethoscope, by dividing the abdomen into four quadrants and evaluating each quadrant. The number of the intestinal sounds in one minute were counted and recorded.
Length of stay in hospital | average of 2 days
  the length of hospital stay (throughout their hospital stay, average of 2 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No